CLINICAL TRIAL: NCT00593580
Title: The Impact of Bisphosphonates on Bone Loss in Patients Undergoing Surgery and Postoperative Chemotherapy for Gynecologic Malignancies.
Brief Title: Bone Health in Gynecologic Cancers-does FOSAVANCE Help?
Acronym: FOSAVANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Jessica McAlpine, MD, UBC and BCCA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H06-03974; 9427-UO146-93C
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; bone mineral density; bisphosphonates; chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Alendronate; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): FOSAVANCE (70 mg/2800 IU of alendronate and cholecalciferol) or placebo will be given weekly for 1 years duration
  Interventions: Drug: alendronate/cholecalciferol
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo
  Arms: 2
Drug: alendronate/cholecalciferol — FOSAVANCE (70 mg/2800 IU of alendronate and cholecalciferol) or placebo will be given weekly for 1 years duration
  Other Names: FOSAVANCE
  Arms: 1

SUMMARY:
Women who undergo bilateral oophorectomy and receive chemotherapy are at risk of increased bone loss. At present, despite having a risk factor profile that fits the indications for assessment and treatment there are no routine interventions in this patient population i.e., the standard treatment is no treatment. We hope to identify whether or not an intervention may be favorable in these women and change the standard of care in this vulnerable population.

Hypothesis:

Weekly therapy with alendronate + vitamin D (FOSAVANCE) will improve bone health as measured by DEXA scans in women with gynecologic malignancies undergoing chemotherapy as compared with patients receiving placebo.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the impact of bisphosphonates on bone mineral density (BMD=primary endpoint) in women with gynecologic malignancies undergoing chemotherapy.
2. To determine if bone loss in women with gynecologic malignancies undergoing chemotherapy is correlated with any of the clinicopathologic parameters gathered in this investigation i.e., race, tumor stage.

Introduction:

Dramatic bone loss in women during the first five years following cessation of ovarian function has been well documented (1). It is estimated that greater than 1.5 million fractures related to osteoporosis (OP) will occur in the US annually (2) and that 33% of women will have sustained hip fractures by age of 90 years(3). With increasing age also comes increasing risk of many cancers, including ovarian, uterine, breast, lung, and colon cancers. 23,500 new cases of ovarian cancer and 38,400 new cases of uterine cancer were diagnosed in the US last year (4). Many of these patients are postmenopausal at the time of diagnosis, and many enter menopause secondary to surgical resection of the ovaries or chemotherapy prompting ovarian failure. This population of women therefore, is at significant risk for osteoporosis.

To the author's knowledge, there has only been one study examining bone loss in menopausal women with gynecologic cancers undergoing chemotherapy (5). This was a small (n=25) prospective observational study with no controlled treatment arm. The authors observed a higher incidence of baseline bone loss and significant additional loss during chemotherapy treatment. Bone loss has also been described in breast cancer patients undergoing chemotherapy (6,7). Laboratory and animal studies demonstrate a deleterious effect of cytotoxic chemotherapy on protein synthesis and DNA replication, resulting in altered or diminished bone formation (8-10). We know of no intervention studies in postmenopausal women with cancer undergoing chemotherapy i.e., comparing different osteoporosis prevention strategies. Estrogen therapy is often contraindicated in gynecologic malignancies and alternative treatments for bone loss prevention are not routinely used by gynecologic oncologists. At present there are no guidelines and/or recommendations in the Gynecologic Oncology community for preventative treatment of bone loss in individuals undergoing chemotherapy (not even calcium and/or vitamin D supplementation recommendations).

Justification:

Women who undergo bilateral oophorectomy and receive chemotherapy are at risk of increased bone loss. At present, despite having a risk factor profile that fits the indications for assessment and treatment there are no routine interventions in this patient population i.e., the standard treatment is no treatment. We hope to identify whether or not an intervention may be favorable in these women and change the standard of care in this vulnerable population.

The use of placebo is justified in this investigation as our current standard of care does not include any treatment for prevention of bone loss during chemotherapy. A recent survey of our patients in active treatment at the BCCA revealed that only 1 of over 40 patients with gynecologic malignancies undergoing chemotherapy was taking any medical therapy for bone loss (Personal communication, J McAlpine J Pike). In order to provide some support for bone mineral density (BMD), all patients enrolled in this study (treatment and control arms) will receive Calcium (1000mg) and Vitamin D supplementation (1000 mg) during the 12 month study period. FOSAVANCE was chosen as the bisphophonate in this investigation as it is the most popular bisphosphonate in Canada and routinely prescribed to thousands of men and women. It has undergone rigorous scrutiny at the federal and provincial levels. Recently, Vitamin D has received considerable press for its "anti-cancer" activity in addition to its known contribution to bone growth and remodeling.

Research Plan:

This is a randomized prospective trial in which women who have undergone surgery for pathology confirmed ovarian (or more rarely advanced stage endometrial) malignancy and scheduled to initiate 6 cycles of chemotherapy (without radiation) will be asked to participate. The primary outcome measured will be change in bone mineral density on consecutive DEXA scans as compared to baseline. All of these patients will have undergone removal of their ovaries bilaterally. Some patients may have entered menopause naturally many years prior to surgical resection of their ovaries. Patients will be told that there will be no difference in their chemotherapy regimen, nor any perceived impact of bisphosphonates on the success of chemotherapy in treating their disease process. Patients fitting the inclusion and exclusion criteria (including blood tests and bone scan criteria) and consenting to participate will be randomized to receive either weekly oral FOSAVANCE 70 mg alendronate/2800 IU cholecalciferol or placebo for the 12 months of the study duration. All patients will receive calcium 1000 mg and vitamin D supplementation 1000 IU daily throughout the study period. Bone DEXA scans will be obtained at baseline (post-surgery and prior to initiation of chemotherapeutic regimen), and after 6 and 12 months of treatment and comparisons made between BMD in the treatment vs. placebo groups. The use of placebo is justified in this investigation as our current standard of care does not include any treatment for prevention of bone loss during chemotherapy. Internationally, there is no recommendation in our subspecialty to do so.

The following parameters will be collected on the enrolled patients: Age, race, tobacco/smoking history, height/weight/BMI, chemotherapeutic regimen, past medical history, tumor stage, grade, histology, complications, blood loss, length of hospital stay, 24 hour creatinine clearance, and serum albumin.

In addition, , family history of osteoporosis and/or spinal or hip fractures, blood sampling for alkaline phosphatase, calcium and 25(OH)vitamin D levels and a DEXA scan (bone scan) at 0, 6, and 12 months with bone mineral density (BMD) measurements of lumbar spine, left hip, and femoral neck (T and Z-scores) will be obtained. These parameters are of specific interest as they relate to the patients bone health and risk factors for bone loss. DEXA scans of individual patients at 6 and 12 months will be compared to their starting/baseline DEXA, and the differences in measurements then compared between patients in the treatment vs. placebo arms. Careful monitoring of patients subjective complaints/comments, complete physical examinations, and monthly laboratory work will be closely monitored throughout the study period.

NOTE: THERE IS NO INTERVENTION IN THIS INVESTIGATION THAT ALTERS THE POSTOPERATIVE CARE, CLINIC VISITS, CHEMOTHERAPY REGIMEN OR DURATION OF TREATMENT IN THESE PATIENTS AS COMPARED TO OUR STANDARD OF CARE. Patients are free to remove themselves from the study at any time with no compromise to their management.

Inclusion Criteria:

1. Postmenopausal (surgical extirpation of ovaries)
2. Primary ovarian or endometrial cancer
3. Planned to receive multiagent chemotherapeutic regimen for 6 cycles
4. Signed informed consent
5. BMD T-score between -2.5 and 0 at any site

Exclusion criteria:

1. Renal insufficiency with CrCl < 35mL/min
2. BMD T-score < -2.5 at any site
3. Medication, excessive alcohol intake, or GI disease inhibiting GI absorption
4. Metabolic bone disease, bony metastases, poorly controlled thyroid or parathyroid conditions, Paget's disease, or on hormonal therapy/other treatments for OP
5. Abnormalities of the esophagus which delay esophageal emptying i.e., achalasia
6. Inability to stand or sit upright for at least 30 minutes
7. Hypersensitivity to any component of the drug product
8. Requiring/planned external beam radiation during study period
9. Baseline serum 25(OH) vitamin D levels of < 9ng/mL

Recruitment:

All patients recruited for this study come from the Gynecologic Oncology clinic via referrals/consultations and are patients of the primary and co-investigators in this study. Prior to enrollment, the investigators will have pathology results and will have made a decision as to whether or not patients require further chemotherapy for their disease process. If the basic inclusion and exclusion criteria are met by demographic/medical/pathology parameters and the patient is interested and has consented for the study, the additional blood work and bone scan will be obtained to ensure that all criteria have been met. All investigators and support staff will be available to review the protocol in detail with patients and phone numbers given to call us with any additional questions.

There is no research nurse or BCCA resources used for this protocol. All discussion of the consent will be done by the PI or one of the Co-investigators. Labs outside of routine BCCA orders (i.e., vitamin D levels) will be done at an outside facility as will DEXA scans and data analysis. Drug/placebo will be delivered by the principal investigator and no pharmacy services are required.

Statistical Analysis:

This is a project looking to detect a 2-3% difference in BMD on DEXA scans as compared to the individuals' baseline DEXA. Based on previous data 11 and our own power analysis this will be achievable with a sample size of 30 patients in each arm (treatment vs. placebo) to ensure sufficient power (Kalloger Consulting, Inc). Our initial analysis will be performed after 30 patients have been randomized (15 FOSAVANCE, 15 placebo). Iif a clear advantage is demonstrated in the treatment group, the trial will be completed and treatment will be offered to all patients undergoing chemotherapy for gynecologic malignancies. If the difference is not yet statistically significant but a favorable trend is suggested we will enroll further patients in order to sufficiently power this series, again with the above specified goal of detecting a 2-3% difference in BMD, considered of clinical signficiance in the literature.

Multiple parameters will be collected (outlined page 2) for descriptive statistics and bivariate analysis, testing for an association of osteoporosis and clinicopathologic and laboratory risk factors. These will be compared between the treatment and control arms to ensure both groups are representative and without potential confounding variables. Paired t-tests will be performed using statistical software (SAS) for the comparison of baseline, 6 and 12-month BMD values, with a significance level of 0.05 and a power of 0.80.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal (surgical extirpation of ovaries)
2. Primary ovarian or endometrial cancer
3. Planned to receive multiagent chemotherapeutic regimen for 6 cycles
4. Signed informed consent
5. BMD T-score between -2.5 and 0 at any site

Exclusion Criteria:

1. Renal insufficiency with CrCl < 35mL/min
2. BMD T-score < -2.5 at any site
3. Medication, excessive alcohol intake, or GI disease inhibiting GI absorption
4. Metabolic bone disease, bony metastases, poorly controlled thyroid or parathyroid conditions, Paget's disease, or on hormonal therapy/other treatments for OP
5. Abnormalities of the esophagus which delay esophageal emptying i.e., achalasia
6. Inability to stand or sit upright for at least 30 minutes
7. Hypersensitivity to any component of the drug product
8. Requiring/planned external beam radiation during study period
9. Baseline serum 25(OH) vitamin D levels of < 9ng/mL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica McALpine, MD, Principal Investigator — UBC/BCCA
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada